CLINICAL TRIAL: NCT04003467
Title: A Six-month Phase 2 Study of Oral hPTH(1-34) (EBP05) in Postmenopausal Women With Low Bone Mass
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Entera Bio Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENT-07-2019
Record Dates: First submitted 2019-06-25; First posted 2019-07-01 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; hPTH(1-34)
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- EBP05 1.5mg (Experimental): subjects will be randomly assigned to receive 3 tablets of EBP05 containing 0.5mg hPTH(1-34) orally each day for 6 months
  Interventions: Drug: EBP05
- Placebo for EBP05 0.5mg (1, 2, 3 or 5) (Experimental): subjects will be randomly assigned to receive 3 or 5 tablets of matching EBP05 placebo orally each day for 6 months
  Interventions: Drug: Placebo of EBP05
- EBP05 2.5mg (Experimental): subjects will be randomly assigned to receive 5 tablets of EBP05 containing 0.5mg hPTH(1-34) orally each day for 6 months
  Interventions: Drug: EBP05
- EBP05 0.5mg (Experimental): subjects will be randomly assigned to receive 1 tablet of EBP05 containing 0.5mg hPTH(1-34) orally each day for 6 months
  Interventions: Drug: EBP05
- EBP05 1.0mg (Experimental): subjects will be randomly assigned to receive 2 tablets of EBP05 containing 0.5mg hPTH(1-34) orally each day for 6 months
  Interventions: Drug: EBP05

INTERVENTIONS:
Drug: EBP05 — tablets
  Other Names: hPTH(1-34); Teriparatide
  Arms: EBP05 0.5mg; EBP05 1.0mg; EBP05 1.5mg; EBP05 2.5mg
Drug: Placebo of EBP05 — tablets
  Other Names: Placebo
  Arms: Placebo for EBP05 0.5mg (1, 2, 3 or 5)

SUMMARY:
This is a double-blinded randomized study to determine the effects of treatment on biochemical markers of bone formation and bone resorption, and bone mineral density (BMD) for 6 months of treatment with EBP05 or placebo. Approximately 160 postmenopausal women with low bone mass (BMD T-score lower than or equal to -2.0 in at least one location: Lumbar Spine, Femoral Neck or Total Hip sites) over 50 years of age will receive Study Medication. Protocol Version 3.0 describes the treatment and evaluation of the initial 103 subjects randomized. In Protocol Version 4.0 the treatment phase will consist of 4 different treatment arms as follows:

Oral EBP05 0.5mg x3 tablets (1.5mg), N=6 Oral EBP05 0.5mg x5 tablets (2.5mg), N=36 Oral Placebo for EBP05 0.5mg (split to sub-groups of: 3 or 5 tablets), N=18

DETAILED DESCRIPTION:
This is a double-blinded randomized study to determine the effects of treatment on biochemical markers of bone formation and bone resorption after 6 months of treatment with EBP05 or placebo. Approximately 160 postmenopausal women with low bone mass (BMD T-score less than or equal to -2.0 in at least one location: Lumbar Spine, Femoral Neck or Total Hip sites) over 50 years of age will be enrolled.

Protocol Version 3.0 described the study design for the initial 103 subjects randomized. The current Version 4.0 describes the study design for approximately 60 additional randomized subjects.

The screening phase to evaluate subject eligibility may start 56 days prior to the treatment phase. BMD screening (DXA scan) will be performed locally on approved vendors standardized machines and interpreted locally. If a subject is found to be suitable, the BMD results will be sent for central reading. The screening DXA scan should be sent to the central reading vendor at least 10 days prior to scheduled potential Day 1 in order to allow timely turnaround of results. The site will receive unblinded results.

A DXA BMD scan performed for medical care unrelated to the study may be used as the screening BMD if obtained no more than 14 days prior the start of screening and performed with the same scanner which was qualified for the study and according to the study specific guidelines and procedures referenced in section 8.1.2. If the subject is eligible for randomization, the DXA scan does not have to be repeated unless there is a delay in the start of Study Medication beyond the 28-day Screening period (see 4.4.3, Extension of Screening window).

Protocol Version 3.0 describes the randomization of the first 103 subjects. In Protocol version 4.0, after completion of all screening procedures eligible subjects will come for the first visit and will be randomized to one of three treatment arms (EBP05 1.5 mg, 2.5 mg or placebo). A randomized allocation schedule will allocate 6 to EBP05 1.5 mg, 36 to 2.5 mg and 18 to placebo.

In Protocol Version 5.0 the starting dose of EBP05 for subjects randomized into the EBP05 2.5 mg treatment group was changed to 1.5 mg (3 tablets). Subjects randomized to Placebo and assigned to the 5 placebo tablet group will also be started on 3 tablets. At the Month 1 visit, the starting dose will be increased to 4 tablets of EPB05 (2.0 mg) or placebo if no continuing drug-related AEs (as assessed by the Investiagor) are present. At Month 2 the dose will be increased to 5 tablets of EPB05 (2.5 mg) or placebo if no continuing drug-related AEs are present. If symptoms associated with administration of Study Medication occur with a dose increase, the dose should be decreased to 3 tablets daily (1.5 mg). Subjects who tolerate the highest dose (5 tablets ,2.5 mg) without drug-related sympoms will continue on that dose for the remainder of the study. Subjects who do not tolerate a dose increase (either 3 tablets to 4 tablets or 4 tablets to 5 tablets) will have their dose reduced to 3 tablets (1.5 mg) daily.

Subjects will receive Study Medication and education on Study Medication intake.

Subjects will visit the clinic once a month for the first three months, and at 6 months for the end of treatment or at any time in-between for an Early Termination Visit, if applicable. There will be telephone calls at Week 2, Month 4 and Month 5 for a general compliance/safety check. The final follow-up visit will also be conducted by phone.

The 6-month DXA scan will be sent for central reading. Unblinded results will not be released to the sites prior to Data Base Lock.

At the End of Treatment visit, concomitant medications will be reviewed, and outcome of AEs recorded, if applicable. The subjects must return all used Study Medication containers. Unused medication should also be returned, collected and accounted for.

ELIGIBILITY:
Inclusion criteria:

1. Female subjects above 50 years of age
2. Signed Informed Consent Form
3. Able to adhere to the visit schedule and protocol requirements
4. At least 3 years post menopause (physiological or surgical)
5. Women who are less than 55 years old need to have estradiol and LH in the menopausal range
6. Low bone mass (BMD T-score lower than or equal to -2.0 in at least one location: Lumbar Spine, Femoral Neck or Total Hip sites)

   Exclusion criteria:
7. Active gastrointestinal inflammatory disorder, gastrointestinal motility disorders, and chronic gastritis, such as ulcerative colitis, Crohn's disease, irritable bowel syndrome, short bowel syndrome, celiac disease, gastroparesis, etc. that may affect drug bioavailability
8. Any conditions or factors that, in the judgment of the Investigator, somehow may impact gastrointestinal absorption, distribution or metabolism of parathyroid hormone analogues, or known to potentiate or predispose to undesired effects
9. History of significant gastrointestinal, liver or kidney disease, or surgery (including bariatric surgery) that may affect drug bioavailability
10. Acute illness within 14 days of screening
11. History of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder, that may result in either increased risk or limit her ability to comply with Study Medication administration and scheduled clinical evaluations, as judged by the investigator
12. Blood donation (greater than or equal to 500 mL) within 30 days prior to screening
13. History of Paget's disease of bone
14. History of prior external beam or implant radiation therapy involving the skeleton
15. Active urolithiasis
16. Primary hyperparathyroidism
17. History of alcohol or substance abuse within 3 years prior to screening
18. The subject has used an investigational drug within 30 days before the screening visit
19. Any past treatment with Forteo®
20. History of oncologic disease except for past medical history of a) basal cell or squamous cell skin cancer resected for cure or b) papillary or follicular thyroid cancer localized to the thyroid and resected for cure with no evidence of local or distant recurrence ≥ 5 years after surgery.
21. Allergy to soy or known hypersensitivity to PTH
22. Known allergies or sensitivities to components of the Study Medication
23. Abnormal calcium, magnesium, phosphate or alkaline phosphatase (outside of lab reference ranges and clinically significant) on screening visit
24. Significant renal impairment (eGFR <45mL/min/1.73 m2 as measured by MDRD)
25. Any other clinically significant abnormal biochemistry, hematology or urinalysis at screening that are not explained by a disease recorded in the subject's medical history, as judged by the investigator
26. Chronic morning medication that cannot be taken at least 1-hr post-Study Medication dose
27. Any osteoporosis treatment within the last 2 years. Hormone therapy with oral, transdermal or injectable estradiol, estrogen analog or SERM (e.g. raloxifene) is considered an osteoporosis treatment. Topical estrogen for menopausal vaginal symptoms is permitted.
28. Any use of fluoride (dose greater than 1 mg/day) or strontium ranelate
29. Any use of intravenous bisphosphonate in the last 10 years.
30. Any use of denosumab within the last 3 years
31. Any oral bisphosphonate use for more than 6 months (or Risedronate for over 1 year) in the last 5 years.
32. Any oral bisphosphonate except risedronate for more than 3 years ending in the last 5 years; or risedronate for more than 5 years ending in the last 5 years.
33. Systemic glucocorticoids (current use: ≥ 2.5 mg prednisone or equivalent), or prior use ≥ 5 mg per day for more than 1 week in the last year
34. Hyperthyroidism or hypothyroidism not treated with thyroxine replacement to achieve normal TSH
35. Serious medical conditions currently under evaluation or treatment
36. Disorders of bone and mineral metabolism other than osteoporosis, including a known history of Vitamin D deficiency with metabolic significance that has not been treated with Vitamin D for at least 6 months.
37. Severe osteoporosis defined as a BMD below -3.5 or previous osteoporotic (low-energy trauma) fracture(s) that in the investigator's opinion preclude the use of placebo.
38. The Investigator should exclude subjects at his own judgement, who are at very high risk of osteoporotic fracture(s) and require immediate treatment.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — postmenopausal women with low bone mass
Enrollment: 161 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Mean % change in P1NP from baseline after 3 months of treatment | baseline, 3 months
  Determine the change in P1NP from baseline during treatment with oral EBP05 for 3 months compared with the change during treatment with placebo

SECONDARY OUTCOMES:
Mean % change in BMD (lumbar) from baseline after 6 months of treatment | baseline, 6 months
  Determine the change in BMD (lumbar spine) from Baseline at Month 6 compared with the change during treatment with placebo
Mean % change in BMD (Femoral Neck and Total Hip) from baseline after 6 months of treatment | baseline, 6 months
  Determine the change in BMD (Femoral Neck and Total Hip) from Baseline at Month 6 compared with the change during treatment with placebo.
Mean % change in P1NP from baseline after 6 months of treatment | baseline, 6 months
  Determine the change in P1NP from baseline during treatment with oral EBP05 for 6 months compared with the change during treatment with placebo.
Mean % change in osteocalcin and bone alkaline phosphatase from baseline after 6 months of treatment | baseline, 6 months
  Determine the changes in osteocalcin and bone alkaline phosphatase from baseline during treatment with oral EBP05 for 3 and 6 months compared with the change during treatment with placebo.
Mean % change in serum CTX and urine NTX/Creatinine from baseline after 3 months of treatment | baseline, 3 months
  Determine the change in serum CTX and urine NTX/Creatinine from baseline during treatment with oral EBP05 for 3 months compared with the change during treatment with placebo.
Mean % change in serum CTX and urine NTX/Creatinine from baseline after 6 months of treatment Change of BMD (lumbar) after 6 months of treatment | baseline, 6 months
  Determine the changes in serum CTX and urine NTX/Creatinine from baseline during treatment with oral EBP05 for 6 months compared with the change during treatment with placebo.
Concentration of plasma hPTH(1-34) 15 min after Study Medication administration | 6 months
  Provide descriptive statistics of plasma hPTH(1-34) concentration 15 min. after Study Medication administration at Day 1, Month 1, Month 3 and Month 6 by treatment group

OTHER OUTCOMES:
Mean % change in urine cyclic AMP/ creatinine by treatment groups | 6 months
  Determine the effect of treatment with EBP05 and placebo on urine cyclic AMP/ creatinine (total urine collected over 1.5-hour post dose) on Day 1, Month 1, Month 3 and Month 6 as a pharmacodynamic response to EPB05
Correlation between mean urine cyclic AMP/ creatinine at Month 3 and Month 6 and mean % change in P1NP from baseline at Months 3 and 6 | 6 months
  Evaluate the correlation between urine cyclic AMP/ creatinine (total urine collected over 1.5-hour post dose) at Month 3 and Month 6 and P1NP change from baseline at Months 3 and 6
Correlation between plasma hPTH(1-34) and urine cyclic AMP/ creatinine at different timepoints | 6 months
  Evaluate the correlation between plasma hPTH(1-34) 15 minutes after oral administration of EBP05 and urine cyclic AMP/ creatinine (total urine collected over 1.5-hour post dose).

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Santora, MD, Study Director — Entera Bio Ltd.
Locations (4):
- Israel (4):
  - Hadassah Medical Center, Mt. Scopus Hospital, Jerusalem
  - Rabin Medical Center, Beilinson Campus, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No